CLINICAL TRIAL: NCT06958601
Title: Comparative Analysis of the Safety and Efficacy of Transoral Robotic Thyroidectomy Versus Conventional Open Thyroidectomy
Brief Title: Safety and Efficacy of Transoral Robotic Thyroidectomy Versus Traditional Open Thyroidectomy for Thyroid Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: No.357[2024]
Record Dates: First submitted 2025-04-06; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Thyroid Cancers
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- traditional open group: 1) General demographic information: including age, gender, ethnicity, etc. 2) Disease-related information: lesion size, lesion location, pathological type, parathyroid function (preoperative, first day postoperative, and one week postoperative), thyroid function (preoperative and one month postoperative), etc.3) Surgery-related information: occurrence of postoperative complications, total number of days of hospitalization following the operation, postoperative quality of life (dysphagia index, neck injury index), etc.
  Interventions: Other: surgical procedure
- robotic group: 1) General demographic information: including age, gender, ethnicity, etc. 2) Disease-related information: lesion size, lesion location, pathological type, parathyroid function (preoperative, first day postoperative, and one week postoperative), thyroid function (preoperative and one month postoperative), etc.3) Surgery-related information: occurrence of postoperative complications, total number of days of hospitalization following the operation, postoperative quality of life (dysphagia index, neck injury index), etc.

INTERVENTIONS:
Other: surgical procedure — Effectiveness of different surgical modalities in the treatment of thyroid cancer
  Groups: traditional open group

SUMMARY:
In general, the utilization of the transoral vestibular approach in robotic surgery demonstrates efficacy comparable to that of traditional open surgery in the treatment of thyroid cancer. This method not only reduces the length of hospitalization for patients but also ensures superior cosmetic outcomes in the cervical region, thus achieving truly scarless aesthetics. The feasibility of Transoral Vestibular Robotic Thyroidectomy (TOVRT) for tumors greater than 2 cm in diameter warrants further exploration in future studies; however, for tumors less than 2 cm in diameter, TOVRT emerges as a safe, reliable, and practical alternative, poised to establish itself as an innovative surgical modality.

ELIGIBILITY:
Inclusion Criteria:

* Age 18- 65 years old, both male and female
* Postoperative pathology was papillary thyroid carcinoma
* Clinical data integrity

Exclusion Criteria:

* Postoperative pathology was benign
* Clinical data are incomplete

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thyroid cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Key Observational Indicators | 6moths
  Incidental parathyroidectomy rate

SECONDARY OUTCOMES:
Secondary observations | 6months
  Incidence of hypoparathyroidism

OTHER OUTCOMES:
Other Pre-Specified Outcome | 6moths
  Number of lymph nodes cleared

IPD SHARING:
Plan to Share IPD: No